CLINICAL TRIAL: NCT03477695
Title: Improving Posture in Parkinson's Patients Through Home-based Training and Biofeedback
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASMC-17-NG-0728-CTIL
Record Dates: First submitted 2018-03-20; First posted 2018-03-26 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-03

CONDITIONS: Parkinson's Disease and Parkinsonism; Postural Kyphosis
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Upright device (Experimental): Ambulatory use of the Upright device
  Interventions: Device: ambulatory use of the Upright device

INTERVENTIONS:
Device: ambulatory use of the Upright device — Patients will wear the UpRight for a period of two month

SUMMARY:
A stooped posture is one of the characteristic motor symptoms of patients with Parkinson's disease, and has been linked to impairments in ADL and QOL. We aimed to test the efficacy, safety, practical utility and user-friendliness of a posture correction and vibrotactile trunk angle feedback device (the UpRight) in the home setting of patients with Parkinson's disease with a stooped posture.

DETAILED DESCRIPTION:
The subjects will be asked to arrive at the Gait laboratory for Mobility Research at Tel Aviv Medical Center. After a detailed explanation of the research procedure and after signing the consent form, they will be introduced to the UPRIGHT GO device. Participances will practice operating and placing the device on the body.

With the device attached to upper back, a number of short clinical tests will be performed:

1. Complete demographic questionnaires and medical history
2. Walking tests and balance:

   1. Short walks at a comfortable speed with or without dual task.
   2. Stairs
   3. Performing daily tasks, such as entering and exiting a room, negotiating obstacles (shoebox), walking between obstacles, buttons, tying laces, carrying small objects on a tray, bringing a glass of water etc.
   4. Timed "Get up and go test" All tests are supervised by a physiotherapist .

Upon completion of the tests, the UPRIGHT device will be delivered for use and exercise for 2 months. Physiotherapist will guide to maintain the devices (such as charging devices and connecting to power).

At the end of the training period, the participans will be invited again to Gait Lab for post tests.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of Parkinson's disease, as defined in the UK Brain Bank criteria
2. Hoehn and Yahr stage I-III
3. Participants who are at stable medication regimen
4. Able to walk independently for at least 5 minutes with or without support of accessory device.

Exclusion criteria:

1. Mini Mental State Exam (MMSE) score< 24

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Average trunk angle in the sagittal plane using a Postural Analysis Chart | 8 weeks
  Postural Analysis

SECONDARY OUTCOMES:
Patient satisfaction by VAS scores | 8 weeks
  Results for the VAS scores with possible range 0 (worst) to 10 (best)

CONTACTS AND LOCATIONS:
Overall Officials: Nir Giladi, MD, Principal Investigator — TASMC
Locations (1):
- Laboratory for gait and neurodynamics, Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] van Wegen EEH, de Goede CJT, Kwakkel G, van Kordelaar J. Sensor assisted self-management in Parkinson's disease: A feasibility study of ambulatory posture detection and feedback to treat stooped posture. Parkinsonism Relat Disord. 2018 Jan;46 Suppl 1:S57-S61. doi: 10.1016/j.parkreldis.2017.07.024. Epub 2017 Jul 25. PMID 28802759